CLINICAL TRIAL: NCT01221025
Title: Effects of Parecoxib on Emergence Delirium and Postoperative Pain in Elderly Patients Undergoing Abdominal Surgery After General Anesthesia
Brief Title: Effect Study of Parecoxib to Treat Emergence Delirium and Postoperative Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Haihua Shu, The First Affliated Hospital of Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHHparecoxib1
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2010-10

CONDITIONS: Emergence Delirium; Postoperative Pain
Keywords: Parecoxib;; emergence delirium;; postoperative pain;; elderly patients;; abdominal surgery; Parecoxib on emergence agitation and postoperative pain
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative | interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- parecoxib (Experimental): Parecoxib, a water-soluble prodrug of valdecoxib, is a high-selective COX-2 inhibitor that is first available for intravenous administration.
  Interventions: Drug: Parecoxib

INTERVENTIONS:
Drug: Parecoxib — The study group will receive first dose of intravenous (IV) injection of parecoxib sodium 40 mg (in a volume of 2 ml) 60 min before the anticipated end of surgery, followed 2 ml IV injection of parecoxib 40 mg will be occurred at 12, 24 and 36 h after the first dose of parecoxib.
  Other Names: Brand name: Dynastat

SUMMARY:
This prospective, double blind, placebo-controlled, parallel group study will be conducted in three study centers in Guangzhou, China. Patients aged older than 65 (ASA I-III) undergoing primary elective abdominal surgery with general anesthesia will be involved in this study. According to previous studies and our pilot trial, the sample size was estimated to be 900 subjects (each center recruiting 300 patients). All eligible patients will be randomly assigned to one of two groups: study group receiving parecoxib and control group receiving normal saline. All patients will be managed with by a standard clinical anesthesia protocol with a sevoflurane-based general anesthesia with continuous intravenous remifentanil, followed by a postoperative PCA with morphine. The emergence delirium will be evaluated by two persons blinding to medication and grouping using Riker sedation-agitation scale immediately since tracheal extubation and at specific time points until patients being discharged from PACU. Pain intensity assessments and pain relief assessments will also be conducted by the patients at given time points in 2 days postoperatively. The morphine-sparing effect, tolerability and safety of parecoxib will be investigated as well.

DETAILED DESCRIPTION:
The inclusion criteria of this study includes:

* Aged older than 65;
* Primary elective abdominal surgery under general anesthesia;
* Ability to understand how to use pain assessment scales and PCA device.

The outcome measures of this study includes:

* Emergence Delirium Assessment;
* Pain intensity and pain relief efficacy endpoints;
* Tolerability and Safety Assessments

ELIGIBILITY:
Inclusion Criteria:

* Aged older than 65;
* Body weight of at least 50 kg;
* Primary elective abdominal surgery under general anesthesia;
* Preoperative health graded as class ASA I-III, based on medical history and physical examination;
* Ability to understand how to use pain assessment scales and PCA device

Exclusion Criteria:

* Emergency or revised abdominal surgery;
* History of known use of analgesics or any other agent that could interfere with analgesic responses during the up to 24 h before receipt of the study medication which including NSAIDs, tricyclic antidepressants, neuroleptic or antipsychotic agents, or corticosteroids (except routine preoperative medication);
* History of known or suspected drug abuse;
* Known allergy, sensitivity, or contraindication to opioid and non-opioid analgesic drugs;
* History of bleeding disorders, peptic ulceration, or anticoagulant use within the past month;
* History of asthma or bronchospasm;
* History of inflammatory bowel disease, a chronic or acute renal or hepatic disorder, coronary heart disease;
* History of dementia and psychological disorder;
* Contraindication to parecoxib.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
emergence agitation | 45 min after anesthesia
  the incidence of emergence agitation after recovery from general anesthesia before discharging from PACU

SECONDARY OUTCOMES:
The amount of morphine consumption and Pain intensity | 48h postoperatively
  The amount of morphine consumption from PCA pump at PACU, 12, 24, 36, and 48h after first dose of study medication; Pain intensity (NRS scores) at 2, 4, 6, 9, 12, 18, 24, 36 and 48 h after the first dose of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Haihua Shu, MD; Ph D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China